CLINICAL TRIAL: NCT01104870
Title: A 12-Week, Randomized, Dose Response Study of UT-15C (Treprostinil Diethanolamine) SR in Patients With Exercise-Induced Pulmonary Hypertension
Brief Title: A Dose Response Study of UT-15C SR in Patients With Exercise-Induced Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDE-PH-202
Record Dates: First submitted 2010-01-04; First posted 2010-04-16 (Estimated); Results first posted 2015-12-30 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Group 1 (Active Comparator): UT-15C 0.25 mg twice daily
  Interventions: Drug: UT-15C
- Dose Group 2 (Active Comparator): UT-15C 1.25 mg twice daily
  Interventions: Drug: UT-15C
- Dose Group 3 (Active Comparator): UT-15C individual Maximum Tolerated Dose
  Interventions: Drug: UT-15C

INTERVENTIONS:
Drug: UT-15C — oral
  Other Names: treprostinil diethanolamine, sustained release

SUMMARY:
This is a prospective, randomized, parallel group study to assess the hemodynamic effect of three different dose regimens of a sustained release (SR) tablet of UT-15C in patients with exercise-induced pulmonary hypertension (PH), as measured by the change in peak total pulmonary resistance index (TPRI) during exercise from Baseline to Week 12.

DETAILED DESCRIPTION:
Prospective, randomized, parallel group study with two periods: a 10 week, dose titration period, followed by a 2 week, dose maintenance period in patients with exercise-induced PH.

The study population will be randomized into Dose Group 1, Dose Group 2, or an Individual Maximum Tolerated Dose (iMTD) of UT-15C SR by Week 10 and maintained through Week 12. Patients may be either currently receiving an approved oral background therapy for their PH (phosphodiesterase-5 [PDE-5] inhibitor, OR endothelin receptor antagonist [ERA]) (no dual background therapy), or not currently receiving therapy for PH.

ELIGIBILITY:
Inclusion Criteria-

A subject was eligible for inclusion in this study if all of the following criteria applied:

1. Was between the ages of 18 and 75 years of age at Screening
2. Weighed a minimum of 40 kilograms with a body mass index less than 40 kg/m2 at Screening
3. Agreed to have right heart catheterization with exercise performed at Baseline and Week 12, or at the time of early discontinuation of study drug
4. Had exercise-induced PH at Baseline (defined as a PAPm ≥ 30 mmHg during exercise).

   Note: eligible subjects may or may not have had a PAPm ≥ 25 mmHg at rest
5. Exercise-induced PH may have been:

   1. Idiopathic, heritable, drug- or toxin-induced PAH, or PAH associated with connective tissue diseases or HIV infection
   2. Due to ILD
   3. Due to sarcoidosis
6. Had a Baseline pulmonary function tests as follows:

   1. Forced vital capacity (FVC) ≥ 50% (predicted)
   2. If FVC <50% (predicted), total lung capacity (TLC) must be ≥ 50% (predicted)
   3. Forced expiratory volume / forced vital capacity (FEV / FVC) ratio ≥ 50%
7. Had a Baseline 6MWD between 150 and 450 meters, inclusive
8. Was optimally treated with conventional pulmonary hypertension therapy (e.g. oral vasodilators, oxygen, digoxin, etc) with no additions, discontinuations, or dose changes for at least 14 days prior to Baseline (excluding anticoagulants). Oral diuretics may have been adjusted, but not discontinued or added, within 14 days of Baseline
9. May or may not have been receiving an approved PDE-5 inhibitor OR an approved ERA.

   Subjects receiving an approved ERA or an approved PDE-5 inhibitor must have been on a stable dose for 30 days prior to Baseline, and were willing to remain on a PDE-5 inhibitor or an ERA and at the same dose for the duration of the 12-week Treatment Phase. If a subject chose to discontinue their PDE-5 or ERA prior to entering this study, they must have had a ≥30 day washout period between the last dose of the PDE-5 or ERA and start of the screening phase.
10. If female, was physiologically incapable of childbearing or practicing an acceptable method of birth control as deemed appropriate by the physician or institution. Women of childbearing potential had a negative serum pregnancy test at Screening
11. Was able to communicate effectively with study personnel, and considered reliable, willing and likely to be cooperative with protocol requirements, including attending all study visits, in the opinion of the Principal Investigator
12. Voluntarily gave informed consent to participate in the study.

Exclusion Criteria-

A subject was not eligible for inclusion in this study if any of the following criteria applied:

1. Had received epoprostenol, treprostinil, iloprost, beraprost, or any other prostacyclin therapy within 30 days of Baseline (except if used during acute vasoreactivity testing)
2. Had previous intolerance or significant lack of efficacy to an oral or parenteral prostacyclin or prostacyclin analogue that resulted in discontinuation or inability to effectively titrate that therapy
3. Had a concurrent injury, illness (other than PH or a PH related condition), or other confounding factor that would prevent the accurate assessment of the subject's exercise capacity
4. Had a musculoskeletal disorder (e.g. recent hip replacement, artificial leg, etc.) or any other disease that was likely to limit ambulation, or was connected to a machine that was not portable
5. Had portal hypertension
6. Had congenital heart disease (repaired or unrepaired)
7. Had a history or current evidence of left-sided heart disease including myocardial infarction in the previous 3 years or mitral valve stenosis, or evidence of current left-sided heart disease as defined by mean resting pulmonary capillary wedge pressure (PCWPm) or left ventricular end diastolic pressure (LVEDP) > 15 mmHg or left ventricular ejection fraction (LVEF) < 45% (as assessed by either multigated acquisition [MUGA] scan, angiography or echocardiography), or symptomatic coronary artery disease (i.e., demonstrable ischemia either at rest or during exercise)
8. Had acute pulmonary embolism (less than 6 months), chronic thromboembolic disease, pulmonary veno-occlusive disease, or pulmonary capillary hemangiomatosis
9. Had an atrial septostomy
10. Had a current diagnosis of uncontrolled sleep disordered breathing
11. Had PH associated with:

    1. chronic obstructive lung disease (COPD), cystic fibrosis, emphysema, alveolar hypoventilation disorders, chronic exposure to high altitude, developmental abnormalities, schistosomiasis, or chronic hemolytic anemia
    2. hematologic disorders (myeloproliferative disorders, splenectomy)
    3. metabolic disorders (glycogen storage disease, Gaucher disease, thyroid disorders
    4. pulmonary Langerhans cell histiocytosis, lymphangioleiomyomatosis, neurofibromatosis, vasculitis
    5. tumoral obstruction, fibrosing mediastinitis, or extensive loss of lung tissue from surgery or trauma
12. Had chronic renal insufficiency as defined by either a Screening creatinine value greater than 2.5 mg/dL (221 μmol/L) or the requirement for dialysis.
13. Had liver function tests (AST or ALT) greater than three times the upper limit of normal at Screening.
14. Had anemia as defined by a Screening hemoglobin value of less than 10 g/dL, active infection, or any other condition that would interfere with the interpretation of study assessments.
15. Had uncontrolled systemic hypertension as evidenced by systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg.
16. Was pregnant or nursing.
17. Had an unstable psychiatric condition or was mentally incapable of understanding the objectives, nature, or consequences of the trial, or had any condition which in the Investigator's opinion would constitute an unacceptable risk to the subject's safety.
18. Was receiving an investigational drug, had an investigational device in place or had participated in an investigational drug or device study within 30 days prior to Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajan Saggar, MD, Principal Investigator — UCLA Pulmonary Division
Locations (9):
- United States (9):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California Los Angeles Pulmonary Division, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Rochester Medical Center, Mary Parkes Center, Rochester, New York
  - The Carl and Edyth Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this study was May 2010 to October 2012. Sites were located in the US only.
Pre-assignment Details: The 50 subjects who received a dose of study drug are presented here.
Groups:
- Dose Group 1: 0.25 mg twice daily
  UT-15C: oral
- Dose Group 2: 1.25 mg twice daily
  UT-15C: oral
- Dose Group 3: individual Maximum Tolerated Dose
  UT-15C: oral
Period: Overall Study
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3
Started | 11 | 19 | 20
Completed | 10 | 18 | 18
Not Completed | 1 | 1 | 2
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Total
Number analyzed (Participants) | 11 | 19 | 20 | 50
Age, Continuous [Mean (Full Range); unit: years] | 53.1 [22 to 74] | 58.9 [43 to 75] | 57.6 [32 to 72] | 57.1 [22 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 15 | 41
  Male | 0 | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3 | 6
  Not Hispanic or Latino | 11 | 16 | 17 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 10 | 18 | 19 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 19 | 20 | 50
PAH History [Number; unit: participants]
  Idiopathic, heritable or drug or toxin-induced PAH | 5 | 6 | 6 | 17
  PAH associated with connective tissue diseases | 5 | 9 | 10 | 24
  PAH associated with HIV | 0 | 0 | 0 | 0
  PH associated with interstitial lung disease (ILD) | 0 | 4 | 3 | 7
  PH associated with sarcoidosis | 1 | 0 | 1 | 2
Background PAH Therapy [Number; unit: participants]
  Both PDE-5i and ERA Dual Therapy | 0 | 0 | 1 | 1
  ERA | 4 | 4 | 1 | 9
  PDE-5i | 3 | 6 | 7 | 16
  No Background Therapy | 4 | 9 | 11 | 24
Baseline Six-Minute Walk Distance (6MWD) [Mean (Standard Deviation); unit: meters] | 366.0 (79.6) | 338.1 (55.7) | 311.4 (67.4) | 333.6 (68.1)
World Health Organization (WHO) Functional Class [Number; unit: participants] — Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms.
  participants
    Class I | 0 | 0 | 0 | 0
    Class II | 2 | 5 | 4 | 11
    Class III | 9 | 14 | 16 | 39
    Class IV | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Total Pulmonary Resistance Index (TPRI) During Exercise From Baseline to Week 12
Description: The effects of 12-week treatment with different doses of UT-15C on peak TPRI during exercise will be evaluated by comparing the change from Baseline to Week 12 at peak wattage on a pairwise basis between treatment groups.
  The primary measure of efficacy was the change from Baseline to Week 12 in peak TPRI during exercise assessed 3 to 6 hours after the subject's morning dose of UT-15C to obtain measurements at peak concentrations of treprostinil. The equation used to determine the Total Pulmonary Resistance Index (TPRI) (mmHg/[L/min/m^2]) is Mean Pulmonary Artery Pressure (PAPm)/ Cardiac Index (CI).
Time Frame: Baseline and Week 12
Population: All subjects with Baseline and Week 12 TPRI values recorded were included in the analysis.
Measure: Mean (Standard Deviation); unit: mmHg/(L/min/m^2)
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3
Number analyzed (Participants) | 10 | 14 | 17
mmHg/(L/min/m^2)
  Baseline | 15.096 (11.668) | 13.954 (9.397) | 15.441 (10.013)
  Week 12 | 14.608 (9.274) | 14.509 (9.463) | 13.423 (7.257)
  Change from Baseline | -0.488 (7.132) | 0.555 (4.428) | -2.019 (5.332)
Statistical Analysis 1: Comparison: Dose Group 1 vs Dose Group 2; Peak total pulmonary resistance index (TPRI) is defined as the TPRI value observed during exercise at the highest matching wattage achieved at both Baseline and Week 12. Where peak wattage cannot be matched, the closest higher wattage will be chosen for comparison; Test type: Superiority or Other; p = 0.95, Wilcoxon (Mann-Whitney) — Primary comparisons are between Dose Group 1 & Dose Group 3 and Dose Group 1 & Dose Group 2. The study is not powered to test for a difference between Dose Group 2 & Dose Group 3
Statistical Analysis 2: Comparison: Dose Group 1 vs Dose Group 3; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change in Mean Pulmonary Artery Pressure (PAPm) From Baseline to Week 12
Description: Pulmonary hypertension (PH) is an increase in pressure in the pulmonary vasculature defined as a mean pulmonary artery pressure (PAPm) greater than 25 mmHg at rest or greater than 30 mmHg with exercise, as measured by right heart catheterization. The PAPm values and their respective changes from Baseline to Week 12 at peak exercise will be summarized by treatment group and measured by Swan-Ganz right heart catheterization.
Time Frame: Baseline and Week 12
Population: All subjects with Baseline and Week 12 PAPm values recorded were included in the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3
Number analyzed (Participants) | 10 | 18 | 18
mmHg
  Baseline | 58.5 (20.7) | 49.1 (11.8) | 51.2 (17.5)
  Week 12 | 58.5 (21.6) | 49.4 (13.4) | 50.8 (14.7)
  Change from Baseline | 0.0 (6.0) | 0.3 (5.4) | -0.4 (6.7)

3. Secondary Outcome: Change in Cardiac Index (CI) From Baseline to Week 12
Description: Cardiac Index (CI) relates the cardiac output (CO) from left ventricle to body surface area (BSA), thus relating heart performance to the size of the individual. The CI values and their respective changes from Baseline to Week 12 at peak exercise will be summarized by treatment group and measured by Swan-Ganz right heart catheterization.
Time Frame: Baseline and Week 12
Population: All subjects with Baseline and Week 12 CI values recorded were included in the analysis.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3
Number analyzed (Participants) | 10 | 14 | 17
L/min/m^2
  Baseline | 5.337 (2.870) | 4.366 (1.462) | 3.940 (1.208)
  Week 12 | 5.313 (3.352) | 4.188 (1.399) | 4.352 (1.372)
  Change from Baseline | -0.024 (1.209) | -0.177 (0.716) | 0.412 (0.959)

4. Secondary Outcome: Change in 6-minute Walk Distance (6MWD) From Baseline to Week 12
Description: The intent of the 6MWD test is to evaluate exercise capacity associated with carrying out activities of daily living. Change in 6MWD from Baseline to Week 12, correlates with the current clinical standard for assessing patient functional status in the treatment of PH and is considered an objective measure of patient functional status by the American Thoracic Society (ATS). Subjects were instructed to walk down a corridor at a comfortable speed as far as they could manage for six minutes. Distance <500 meters suggests considerable exercise limitation; Distance 500-800 meters suggests moderate limitation; Distance >800 meters (with no rests) suggests mild or no limitation.
Time Frame: Baseline and Week 12
Population: All subjects with Baseline and Week 12 6MWD values recorded were included in the analysis.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3
Number analyzed (Participants) | 10 | 18 | 17
meters
  Baseline | 361.5 (82.4) | 338.0 (57.3) | 317.8 (55.2)
  Week 12 | 407.6 (98.2) | 356.7 (89.8) | 349.5 (89.8)
  Change from Baseline | 46.1 (74.9) | 18.7 (74.3) | 31.6 (64.9)

5. Secondary Outcome: Change in Borg Dyspnea Score (Following 6MWT) From Baseline to Week 12
Description: The Borg dyspnea score is a 10-point scale rating the maximum level of dyspnea (difficulty in breathing) experienced during the six-minute walk test (6MWT). The Borg dyspnea score was assessed immediately following the 6MWT. Scores ranged from 0 (for no shortness of breath) to 10 (for the greatest shortness of breath ever experienced).
Time Frame: Baseline and Week 12
Population: All subjects with Baseline and Week 12 Borg dyspnea scores recorded were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3
Number analyzed (Participants) | 10 | 18 | 17
score
  Baseline | 3.0 [1.0 to 5.0] | 3.8 [3.0 to 5.0] | 3.0 [2.0 to 6.0]
  Week 12 | 2.5 [1.0 to 5.0] | 3.0 [2.0 to 6.0] | 3.0 [2.0 to 5.0]
  Change from Baseline | 0.5 [-2.0 to 2.0] | 0.0 [-1.5 to 1.0] | 0.0 [-1.5 to 1.0]

6. Secondary Outcome: Change in PH Symptoms From Baseline to Week 12
Description: Symptoms of PH including fatigue, dyspnea, edema, dizziness, syncope, chest pain and orthopnea were assessed and severity grade values (i.e., 0, 1, 2 or 3) for each symptom were assigned for subjects. A severity of 0 indicated no symptoms, the maximum severity was 3, indicating severe symptoms. Median change in symptom severity from Baseline to Week 12 is described.
Time Frame: Change from Baseline at 12 Weeks
Population: All subjects with Baseline and Week 12 values recorded for symptoms of PH were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3
Number analyzed (Participants) | 10 | 18 | 18
units on a scale
  Change in Fatigue Symptoms from Baseline | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0]
  Change in Dyspnea Symptoms from Baseline | -1.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0] | -0.5 [-1.0 to 0.0]
  Change in Edema Symptoms from Baseline | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 1.0] | 0.0 [-1.0 to 0.0]
  Change in Dizziness Symptoms from Baseline | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0]
  Change in Syncope Symptoms from Baseline | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Change in Chest Pain Symptoms from Baseline | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [0.0 to 0.0]
  Change in Orthopnea Symptoms from Baseline | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0]

7. Secondary Outcome: Number of Participants With a Change From Baseline World Health Organization (WHO) Functional Classification at Week 12
Description: The WHO Functional Class of pulmonary hypertension is a physical activity rating scale as follows: Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms. Only participants who experienced a change in WHO functional classification from Baseline to Week 12 are described by class change below; all other participants maintained their Baseline WHO functional classification at Week 12.
Time Frame: Change from Baseline at Week 12
Population: All subjects with Baseline and Week 12 WHO functional classifications recorded were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3
Number analyzed (Participants) | 10 | 18 | 18
participants
  Change from Class II to Class III | 0 | 0 | 1
  Change from Class III to Class I | 1 | 0 | 0
  Change from Class III to Class II | 2 | 1 | 4

8. Secondary Outcome: Change in N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP) Concentrations From Baseline to Week 12
Description: The N-terminal pro-BNP (NT-proBNP) serum concentration was assessed to compare the severity of heart failure at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: All subjects with Baseline and Week 12 NT-proBNP values recorded were included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3
Number analyzed (Participants) | 10 | 15 | 18
pg/mL
  Baseline | 678.7 (1530.0) | 565.4 (960.0) | 1092.1 (1768.9)
  Week 12 | 654.4 (1133.7) | 750.5 (1223.3) | 1571.7 (2808.6)
  Change from Baseline | -24.4 (592.1) | 185.1 (634.9) | 479.6 (2236.9)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the 12 week study, including the screening phase, as well as 30 days post end of study visit.
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/19 | 4/20
Other Adverse Events (participants affected / at risk) | 11/11 | 17/19 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Group 1 (N=11) | Dose Group 2 (N=19) | Dose Group 3 (N=20)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Group 1 (N=11) | Dose Group 2 (N=19) | Dose Group 3 (N=20)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 13 (13)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 7 (9) | 8 (8)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (5) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 10 (10) | 14 (14)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 2 (2)
Anthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 4 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 5 (5)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 5 (5)
Pain (General disorders) | 2 (2) | 0 (0) | 4 (4)
Oedema peripheral (General disorders) | 0 (0) | 2 (3) | 2 (3)
Catheter site haematoma (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic ulcer (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (4)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 9 (9)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Body temperature decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed, except as provided below. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.